CLINICAL TRIAL: NCT04176445
Title: Influence of Body Positioning on Pulmonary Aeration Among Mechanically Ventilated Critical Ill Patients
Brief Title: Body Positioning and Pulmonary Aeration During Mechanical Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was stopped prematurely due to the COVID-19 pandemic
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Hospital Ernesto Dornelles (Other)
Responsible Party: Principal Investigator, Douglas Neves, Principal Investigator, Hospital Moinhos de Vento
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 3.243.829
Record Dates: First submitted 2019-10-19; First posted 2019-11-25 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2019-11

CONDITIONS: Critical Illness
Keywords: Critical Care; Sitting Position; Tilt Table; Ultrasonography
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: at a single day: arm 1: bedside sitting posture followed by orthostatic board at 45º and 60º; arm 2: orthostatic board at 45º, 60º, and 80º followed by bedside sitting posture.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bedside Sitting followed by Orthostatic Board (Other): Bedside sitting posture protocol followed by orthostatic board posture protocol.
  Interventions: Device: Orthostatic board posture; Other: Bedside sitting posture
- Orthostatic Board followed by Bedside Sitting (Other): Orthostatic board posture protocol followed by bedside sitting posture protocol.
  Interventions: Device: Orthostatic board posture; Other: Bedside sitting posture

INTERVENTIONS:
Device: Orthostatic board posture — Patients will be verticalized at at 45º, 60º and 80º using an orthostatic board. The total posture protocol will last 30 minutes
Other: Bedside sitting posture — Patients will be placed at the bedside, with support for the back and upper limbs. They will be kept at 90º of hip and knee flexion and feet supported. The total posture protocol will last 30 minutes.

SUMMARY:
The present randomized crossover clinical trial aims to evaluate the influence of different body postures on pulmonary aeration among mechanically ventilated critically ill patients. Patients admitted to the intensive care unit receiving invasive mechanical ventilation >24 hours, and without contraindications to mobilization, will be randomly assigned to one of two sequences of interventions at a single day: arm 1: bedside sitting posture followed by orthostatic board at 45º and 60º; arm 2: orthostatic board at 45º, 60º and 80º followed by bedside sitting posture. Each postural protocol (bedside sitting posture protocol or orthostatic board posture protocol) will last 30 minutes. A washout window period between 1,5h and 2,5h will be applied between the two postural interventions. The primary outcome is the lung aeration assessed using the Lung Ultrasound Score (LUS) performed by trained evaluators at the end of postural protocol. Secondary outcomes include ventilatory mechanics (static compliance, airway resistance and respiratory work), PaO2/FiO2 ratio, Level of consciousness according to the Richmond Agitation-Sedation Scale (RASS), and adverse events (hypertension, hypotension, tachicardia, bradycardia, tachypnea, bradypnea, decreased level of consciousness, patient distress, fall to knees, invasive device traction or loss, filter hemodialysis clotting or disruption).

ELIGIBILITY:
Inclusion Criteria: 18 years or older; Invasive Mechanical Ventilation > 24 hours; no weaning expectation on screening day for study eligibility; Signature of Informed Consent.

Exclusion Criteria:

* Patients using vasoative drugs (noradrenaline > 0.2mcg/kg/min or sodium nitroprosside > 1mcg/kg/min);
* Increase > 50% in noradrenaline dose in the last 2 hours; since exceeds 0,1 mcg / kg / min in that period;
* Inclusion of norepinephrine in the last 2 hours, with the dose > 0.1mcg/kg/min;
* Heart rate less than 40 beats per min or more than 130 beats per min
* Active myocardial ischaemia;
* Systolic blood pressure more than 200 mmHg,
* Mean arterial blood pressure less than 65 mm Hg or more than 110 mm Hg;
* Arrhythmia
* Intra-aortic balloon
* RASS <-4 ou > +1;
* Intracranial hypertension;
* Patient agitation
* External ventricular drain;
* Neurologic and/or orthopedic conditions that prevented orthostatism
* spinal cord injury) or
* Spinal cord injury and/or risk od instabilitity
* Acute stroke;
* orthopedic fractures in the lower limf
* Inability to walk with- out assistance before acute ICU illness (use of a cane or walkers its not exclusions;
* MRC > 3 MMII;
* Major pressure ulcers in the calcaneal region;
* FiO2 > 60%
* Positive end-epiratory pressure > 10cmH2O;
* Pulse oximetry less than 88%
* Respiratory rate less than 5 breaths per min or more than 40 breaths per min
* Neuromuscular blocking;
* Reserved Prognosis;
* Peritoneostomy;
* Temperature> 38.5 °C;
* Active gastrointestinal blood loss
* Intra-abdominal Hypertension;
* Thrombocytopenia (platelet count <50 000);
* Diarrhea;
* Hyperglycemia, with HGT < 70mg/g
* Intermittent haemodialysis
* Large abdominal surgery
* Continuous Epidural infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Dal Lago, Study Director — Experimental Physiology Laboratory - Universidade Federal de Ciências da Saúde de Porto Alegre (UFCSPA); Regis Gourlart Rosa, Study Director — Intensive Care Unit, Hospital Moinhos de Vento
Locations (2):
- Brazil (2):
  - Hospital Ernesto Dornelles, Porto Alegre
  - Hospital Moinhos de Vento, Porto Alegre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sonpeayung R, Tantisuwat A, Klinsophon T, Thaveeratitham P. Which Body Position Is the Best for Chest Wall Motion in Healthy Adults? A Meta-Analysis. Respir Care. 2018 Nov;63(11):1439-1451. doi: 10.4187/respcare.06344. Epub 2018 Oct 16. PMID 30327334
- [Background] Perme C, Chandrashekar R. Early mobility and walking program for patients in intensive care units: creating a standard of care. Am J Crit Care. 2009 May;18(3):212-21. doi: 10.4037/ajcc2009598. Epub 2009 Feb 20. PMID 19234100
- [Background] Dong ZH, Yu BX, Sun YB, Fang W, Li L. Effects of early rehabilitation therapy on patients with mechanical ventilation. World J Emerg Med. 2014;5(1):48-52. doi: 10.5847/wjem.j.issn.1920-8642.2014.01.008. PMID 25215147
- [Background] Porto EF, Castro AA, Leite JR, Miranda SV, Lancauth A, Kumpel C. Comparative analysis of respiratory systems compliance in three different positioning (lateral, dorsal and sitting) in patients in prolonged invasive mechanical ventilation. Rev Bras Ter Intensiva. 2008 Sep;20(3):213-9. English, Portuguese. PMID 25307087
- [Background] Chang AT, Boots RJ, Hodges PW, Thomas PJ, Paratz JD. Standing with the assistance of a tilt table improves minute ventilation in chronic critically ill patients. Arch Phys Med Rehabil. 2004 Dec;85(12):1972-6. doi: 10.1016/j.apmr.2004.03.024. PMID 15605335
- [Background] Umei N, Atagi K, Okuno H, Usuke S, Otsuka Y, Ujiro A, Shimaoka H. Impact of mobilisation therapy on the haemodynamic and respiratory status of elderly intubated patients in an intensive care unit: A retrospective analysis. Intensive Crit Care Nurs. 2016 Aug;35:16-21. doi: 10.1016/j.iccn.2016.02.001. Epub 2016 Mar 5. PMID 26961919
- [Background] Sustic A, Protic A, Cicvaric T, Zupan Z. The addition of a brief ultrasound examination to clinical assessment increases the ability to confirm placement of double-lumen endotracheal tubes. J Clin Anesth. 2010 Jun;22(4):246-9. doi: 10.1016/j.jclinane.2009.07.010. PMID 20522353
- [Background] Lichtenstein D, Goldstein I, Mourgeon E, Cluzel P, Grenier P, Rouby JJ. Comparative diagnostic performances of auscultation, chest radiography, and lung ultrasonography in acute respiratory distress syndrome. Anesthesiology. 2004 Jan;100(1):9-15. doi: 10.1097/00000542-200401000-00006. PMID 14695718
- [Background] Bouhemad B, Liu ZH, Arbelot C, Zhang M, Ferarri F, Le-Guen M, Girard M, Lu Q, Rouby JJ. Ultrasound assessment of antibiotic-induced pulmonary reaeration in ventilator-associated pneumonia. Crit Care Med. 2010 Jan;38(1):84-92. doi: 10.1097/CCM.0b013e3181b08cdb. PMID 19633538
- [Background] Bouhemad B, Zhang M, Lu Q, Rouby JJ. Clinical review: Bedside lung ultrasound in critical care practice. Crit Care. 2007;11(1):205. doi: 10.1186/cc5668. PMID 17316468
- [Background] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Background] Soummer A, Perbet S, Brisson H, Arbelot C, Constantin JM, Lu Q, Rouby JJ; Lung Ultrasound Study Group. Ultrasound assessment of lung aeration loss during a successful weaning trial predicts postextubation distress*. Crit Care Med. 2012 Jul;40(7):2064-72. doi: 10.1097/CCM.0b013e31824e68ae. PMID 22584759
- [Derived] Neves D, Marques Filho PR, Townsend RDS, Rodrigues CDS, Tagliari L, Madeira LC, Mattioni MF, Camillis MLF, Leaes CGS, Andrade JMS, Robinson CC, Sganzerla D, Drehmer L, Costa DFMD, Machado AS, Rosa RG, Lago PD. Impact of vertical positioning on lung aeration among mechanically ventilated intensive care unit patients: a randomized crossover clinical trial. Crit Care Sci. 2023 Oct-Dec;35(4):367-376. doi: 10.5935/2965-2774.20230069-en. PMID 38265318

RESULTS

PARTICIPANT FLOW:
Groups:
- Bedside Sitting (First Intervention) Followed by Orthostatic Board (Second Intervention): Bedside sitting posture protocol followed by orthostatic board posture protocol.
  Orthostatic board posture: Patients will be verticalized at at 45º, 60º and 80º using an orthostatic board. The total posture protocol will last 30 minutes
  Bedside sitting posture: Patients will be placed at the bedside, with support for the back and upper limbs. They will be kept at 90º of hip and knee flexion and feet supported. The total posture protocol will last 30 minutes.
- Orthostatic Board (First Intervention) Followed by Bedside Sitting (Second Intervention): Orthostatic board posture protocol followed by bedside sitting posture protocol.
  Orthostatic board posture: Patients will be verticalized at at 45º, 60º and 80º using an orthostatic board. The total posture protocol will last 30 minutes
  Bedside sitting posture: Patients will be placed at the bedside, with support for the back and upper limbs. They will be kept at 90º of hip and knee flexion and feet supported. The total posture protocol will last 30 minutes.
Period: Overall Study
Arm/Group | Bedside Sitting (First Intervention) Followed by Orthostatic Board (Second Intervention) | Orthostatic Board (First Intervention) Followed by Bedside Sitting (Second Intervention)
Started | 12 | 7
Completed | 12 | 5
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — change plans weaning after first intervention | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Study participants were randomized to Bedside sitting (first intervention) posture protocol followed by orthostatic board (second intervention) posture protocol or Orthostatic board (first intervention) posture protocol followed by bedside sitting posture (second intervention) protocol.
  Orthostatic board posture: Patients will be verticalized at at 45º, 60º and 80º using an orthostatic board. The total posture protocol will last 30 minutes
  Bedside sitting posture: Patients will be placed at the bedside, with support for the back and upper limbs. They will be kept at 90º of hip and knee flexion and feet supported. The total posture protocol will last 30 minutes.
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 19
Charlson comorbidity index [Mean (Standard Deviation); unit: score] — One point was assigned to: past history of myocardial infarction, heart failure, peripheral vascular disease, cerebrovascular disease, dementia, chronic lung disease, connective tissue disease, peptic ulcer disease, mild liver disease and diabetes. The comorbidities weighted with 2 points were: diabetes with target organ damage, hemiplegia, moderate to severe renal disease, malignant neoplasm, leukaemia and lymphoma. Moderate to severe liver disease was weighted with 3 points and metastatic solid tumour and AIDS (stage C) were weighted with 6 points. higher values = worse. Total score: summed
  score | 3.2 (1.7)
Reason for mechanical ventilation [Count of Participants; unit: Participants]
  Acute respiratory failure | 11
  Hemodynamic instability | 1
  Decreased level of consciousness | 5
  Cardiac arrest | 2
Duration of Invasive Mechanical Ventilation [Mean (Standard Deviation); unit: days] | 4.3 (1.1)
ICU admission type [Count of Participants; unit: Participants]
  Medical | 18
  Surgical | 1
Simplified Acute Physiology Score 3 [Mean (Standard Deviation); unit: score] — The Simplified Acute Physiology Score 3 prognostic system is composed of 20 variables, represented by an acute physiological score and assessment of the previous state, aiming to establish a predictive index of mortality for patients admitted to intensive care units. The lowest value assigned by the score is 0 and the highest is 217 points, with higher values indicating greater severity.
  score | 71.6 (10.8)
Continuous parenteral sedation [Count of Participants; unit: Participants] | 3
Richmond Agitation-Sedation Scale [Mean (Standard Deviation); unit: score] — The Richmond Agitation-Sedation Scale assesses the level of sedation and agitation of a patient under critical care. Its score ranges from +4 to -5, with the highest value ( +4 ) being described as a combative and violent patient, and the lowest value (-5) described as a patient not responding to verbal or physical stimuli.
  score | -4 (1.1)
Mode of mechanical ventilation [Count of Participants; unit: Participants]
  Presure Support Ventilation | 13
  Pressure Control Continuous Mandatory Ventilation | 6

OUTCOME MEASURES:

1. Primary Outcome: Lung Aeration Scores Post Intervention (Verticalization)
Description: Evaluation of lung aeration using the Lung Ultrassound Score. The division landmark it is the anterior and posterior axillary lines, with each region being divided into upper and lower. Thus, six representative zones of each lung are assessed. Normal aeration is represented by the presence of pleural sliding and horizontal A lines, or by at least three vertical B lines, a 0 score is assigned. When a moderate loss of aeration takes place, characterized by multiple B lines, either regularly or irregularly spaced, originating from the pleural line, a score of 1 is assigned. When coalescent B lines are present in several intercostal spaces occupying the whole intercostal space, a score of 2 is assigned to the region. If there is a total loss of lung aeration, as observed in lung consolidation, a score of 3 is assigned. The total LUS score is achieved by summing the 12 regions examined, with its scores ranging from 0 to 36, and the higher the score, the worse lung aeration.
Time Frame: Single day assessment post intervention of the sitting posture (protocol lasts 30 minutes) and post intervention of the standing board (protocol lasts 30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bedside Sitting: Bedside sitting posture: Patients were placed at the bedside, with support for the back and upper limbs. They were kept at 90º of hip and knee flexion and feet supported. The total posture protocol were last 30 minutes.
- Orthostatic Board: Orthostatic board posture: Patients were verticalized at at 45º, 60º and 80º using an orthostatic board. The total posture protocol were last 30 minutes
Arm/Group | Bedside Sitting | Orthostatic Board
Number analyzed (Participants) | 17 | 19
score on a scale | 13.7 (7.6) | 11.0 (8.0)

2. Secondary Outcome: Tidal Volume
Description: Variations in tidal volume according to body position. Tidal volume expresses the value (in ml) that enters and leaves the lungs at each respiratory cycle. Variations extracted directly from the mechanical ventilation monitor. Outcome has no range, neither higher or lower values are considered to be a better or worse outcome
Time Frame: Single day assessment at the end of sitting posture protocol (the protocol lasts 30 minutes) and at the end of orthostatic board protocol (the protocol lasts 30 minutes).
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Bedside Sitting | Orthostatic Board
Number analyzed (Participants) | 17 | 19
ml | 435 [380 to 480] | 436 [396 to 507]

3. Secondary Outcome: Minute Volume
Description: Variations in minute volume according to body position. Minute volume expresses the value (in L/min) that enters and leaves the lungs during one minute. Variations extracted directly from the mechanical ventilation monitor. Outcome has no range, neither higher or lower values are considered to be a better or worse outcome
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: L/min
Arm/Group | Bedside Sitting | Orthostatic Board
Number analyzed (Participants) | 17 | 19
L/min | 11.1 [8.4 to 12.2] | 10.3 [8.7 to 12.5]

4. Secondary Outcome: Number of Professionals for Verticalization
Description: The absolute number of professionals required to perform each the chest verticalization protocols was counted. Outcome has no range, neither higher or lower values are considered to be a better or worse outcome
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: professionals per procedure
Arm/Group | Bedside Sitting | Orthostatic Board
Number analyzed (Participants) | 17 | 19
professionals per procedure | 3 [3 to 3.3] | 3 [3 to 3]

ADVERSE EVENTS:
Time Frame: The evaluations took place in a single moment/day. Possible adverse events were evaluated from randomization to the last assessment of the outcome.
Arm/Group | Bedside Sitting | Orthostatic Board
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 1/17 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bedside Sitting (N=17) | Orthostatic Board (N=19)
Hypontension (Cardiac disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
* First, just over 50% of the sample target was met; however, the early interruption of the study was necessary due to the health reality imposed by the COVID-19 pandemic.
* Second, due to the nature of the interventions, it is not possible to blind the assessments, which may have led to measurement bias and the Hawthorn effect.
* Third, in addition to the small sample, the study was limited to 2 hospitals, which may limit the external validity in other contexts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT04176445/Prot_SAP_000.pdf